CLINICAL TRIAL: NCT06714604
Title: Standard Versus Prolonged Neoadjuvant (Conversion) Chemotherapy to Prolong Survival of Patients With Borderline and Locally Advanced Pancreatic Cancer: a Phase III Randomized Controlled
Brief Title: Standard or Prolonged Neoadjuvant Chemotherapy Before Surgery for BR/LAPC
Acronym: ADVANTAGE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Elena Rangelova, Principal Investigator, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-502117-29-00
Record Dates: First submitted 2023-02-21; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma; Borderline Resectable Pancreatic Carcinoma; Pancreas Cancer; Neoadjuvant Chemotherapy; Surgery; Pancreatectomy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox

STUDY DESIGN:
Intervention Model Description: Randomized controlled two-arm open label phase 3 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard (Active Comparator): 8 cycles of neoadjuvant mFOLFIRINOX or 4 cycles of neoadjuvant gemcitabine-nab-paclitaxel
  Interventions: Drug: FOLFIRINOX or gemcitabine-nab-paclitaxel
- Prolonged (Experimental): 12 cycles of neoadjuvant mFOLFIRINOX or 6 cycles of neoadjuvant gemcitabine-nab-paclitaxel
  Interventions: Drug: FOLFIRINOX or gemcitabine-nab-paclitaxel

INTERVENTIONS:
Drug: FOLFIRINOX or gemcitabine-nab-paclitaxel — 4 months if treatment
  Arms: Standard
Drug: FOLFIRINOX or gemcitabine-nab-paclitaxel — 6 months of treatment
  Arms: Prolonged

SUMMARY:
The goal of this multicenter randomized controlled phase III trial is to compare two durations of neoadjuvant chemotherapy (NAT) with mFOLFIRINOX or gemcitabine-nab-paclitaxel (GnP) before attempt for surgical resection in patients with borderline (BR) and locally advanced pancreatic cancer (LAPC). Patients with histologically confirmed non-metastatic BR/LAPC evaluated to potentially tolerate any of the treatment regimens and pancreatic surgery will be randomized to receive either standard duration NAT with 6 cycles mFOLFIRINOX or 4 cycles GnP or prolonged duration NAT with either 12 cycles mFOLFIRINOX or 6 cycles GnP before attempt for surgical resection, provided there is no evidence of disease progression. The primary objective is to compare the overall survival at 24 months after randomization of all treated patients and among the resected patients with BR/LAPC.

DETAILED DESCRIPTION:
The prognosis of the large majority cancer types has gradually improved over the past decades. Pancreatic cancer (PC) is one of the few exceptions where the 5-year survival still lies under the 10% threshold. Surgery is the only treatment modality that can contribute to long-term survival. However, only about 20% of the patients qualify for surgery since PC often presents as spread disease at the time of diagnosis. Even after curatively intended surgery the prognosis is still dismal, with a 5-year survival of about 20%. Chemotherapy can reduce the risk for recurrence after surgery.

A factor that complicates surgery is the anatomical location of the pancreas. It overlies the large abdominal vessels, which provide blood supply to the liver and the small bowel. Approximately 25% of the patients present at diagnosis with what is labeled as borderline (BR) or locally advanced pancreatic cancer (LAPC). BR and LAPC refer to different degree of tumoral involvement of the large abdominal vessels. Previously, resection of tumors with this type of vascular involvement has not been a treatment alternative, since the postoperative complication rate has been unacceptably high and there has not been a potent oncologic treatment to address potential micrometastatic spread. Therefore, the survival of patients with BR/LAPC has for long been almost as short as the survival of patients with spread PC.

The introduction of the potent combination chemotherapy FOLFIRINOX significantly improved the survival of patients with BR/LAPC and metastatic PC compared to the previous standard gemcitabine. Patients with BR/LAPC who could be resected after induction chemotherapy with FOLFIRINOX had furthermore chance for long-term term survival compared to unresected patients. Even other types of combination therapy, such as gemcitabine-nab-paclitaxel, have shown to lead to long-tern survival of patients with BR/LAPC who could be resected after initial chemotherapy.

Generally, the larger the tumor size the higher the risk for vascular invasion, lymph node metastases and elevated CA19-9, all associated with worse prognosis. Neoadjuvant chemotherapy contributes to decreased tumor size, lower probably for lymph node metastases and lower CA19-9. In this way the risk for recurrence decreases while the potential benefit of surgery increases. Theoretically, repeated cycles of chemotherapy under longer period would have the possibility to destroy more cancer cells. In studies it has been shown that the duration of chemotherapy is correlated with better histologic tumor regression and chance for negative lymph nodes. On the contrary, it could also be that longer treatment periods induce resistant cell clones which can reverse the previous beneficial treatment effects and decondition the patients. Often there is a limit to what the patient can tolerate in terms of side effects and general condition.

Since the outcome of technically advanced pancreatic surgery has been shown to correlate with volume, a national level structure has been implemented in Sweden, limiting the surgical treatment of BR/LAPC to two national centers with the intention to increase patient safely and improve postoperative outcome. Regarding the length of preoperative chemotherapy, two alternative regimens have been used by the two centers - either six cycles of modified FOLFIRINOX or four cycles of gemcitabine-nab-paclitaxel. Previously published data confirmed that long-term survival can be achieved by these treatment setups. However, internationally it is more common to apply eight or more cycles of FOLFIRINOX for BR/LAPC. In larger international multicenter studies, showing the efficacy of FOLFIRINOX when used with palliative intent or as adjuvant treatment, the aimed number of treatment cycles has been set to twelve. When gemcitabine-nab-paclitaxel has been intended for the treatment of LAPC, six cycles have been administered.

Both FOLFIRINOX and gemcitabine-nab-paclitaxel are well established treatment alternatives in the neoadjuvant setting for BR/LAPC, however, the most optimal treatment duration is unknown. The purpose of this study is to determine the optimal duration of neoadjuvant treatment for BR/LAPC, in an attempt to increase the number of patients who can be resected, and increase the survival of the resected ones and the whole group of patients with BR/LAPC.

The goal of this multicenter randomized controlled phase III trial is to compare two durations of neoadjuvant chemotherapy (NAT) with mFOLFIRINOX or gemcitabine-nab-paclitaxel (GnP) before attempt for surgical resection in patients with borderline (BR) and locally advanced pancreatic cancer (LAPC). Patients with histologically confirmed non-metastatic BR/LAPC evaluated to potentially tolerate any of the treatment regimens and pancreatic surgery will be randomized to receive either standard duration NAT with 6 cycles mFOLFIRINOX or 4 cycles GnP or prolonged duration NAT with either 12 cycles mFOLFIRINOX or 6 cycles GnP before attempt for surgical resection, provided there is no evidence of disease progression. The primary objective is to compare the overall survival at 24 months after randomization of all treated patients and among the resected patients with BR/LAPC. Furthermore, overall and progression-free survival in the who group and among the resected patients will be compared after 60 months in intention-to-treat and in the per protocol treated cohorts. Furthermore, survival will be compared among patients with BR or LAPC separately and between the groups of BR and LAPC.

ELIGIBILITY:
Inclusion Criteria:

* Borderline or locally advanced pancreatic adenocarcinoma at diagnosis according to National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines, version 1.2022
* Histo- or cytologically confirmed adenocarcinoma (preferably EUS-guided)
* T1-4, Nx, M0 according to AJCC 8th edition
* ECOG 0-1 and considered fit for the planned chemotherapy at the local hospital and surgery at the two national centers for BR/LAPC
* Written informed patient consent

Exclusion Criteria:

* Co-morbidity precluding pancreatic surgery or chemotherapy
* Contraindications to any of the drugs in the proposed treatment regimens
* ECOG ≥2
* Neuropathy ≥ grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE), version 6
* Granulocyte count < 1500 per cubic millimetre (< 1,5 x 109/L)
* Platelet count < 100 000 per cubic millimetre (< 100 x 109/L)
* Serum creatinine > 1.5 UNL (upper limit normal range)
* Albumin <2,5 g/dl (<25 g/L)
* Total bilirubin >3 x ULN
* ASAT (SGOT) and ALAT (SGPT) >2.5 x institutional ULN
* female patients in child-bearing age not using adequate contraception, pregnant or lactating women
* mental or somatic disorders which could possibly interfere with informed consent, compliance or the planned treatments
* previous oncologic treatment for PC within the past 5 years
* participation in other clinical trial with an investigational product during the past 30 days
* Any reason according to the investigator why the patient cannot comply with the protocol or is not suitable to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival of all BR/LAPC patients | 24 months of randomization
  Comparison of overall survival of all enrolled BR/LAPC patients treated with the standard or the prolonged treatment
Overall survival of all resected BR/LAPC patients | 24 months of randomization
  Comparison of overall survival of the resected BR/LAPC patients treated with the standard or the prolonged treatment

SECONDARY OUTCOMES:
Overall survival in intention-to-treat and per protocol treated | 60 months
  Comparison of overall survival of all BR/LAPC patients treated with standard or prolonged treatment in intention-to-treat and in the per protocol treated cohorts
Progression-free survival (PFS) in intention-to-treat and per protocol treated | 60 months
  Comparison of progression-free survival of all BR/LAPC patients treated with standard or prolonged treatment in intention-to-treat and in the per protocol treated cohorts
Overall survival among non-resected BR/LAPC patients | 24 months
  Comparison of overall survival of all non-resected BR/LAPC patients treated with standard or prolonged treatment
Overall and progression-free survival among all and among resected patients with BR in the two arms in ITT | 60 months
  Comparison of overall and progression-free survival of patients with BR treated with standard or prolonged treatment. Comparison in survival will be performed among all enrolled patients and among all resected patients with BR receiving the two treatment durations
Overall and progression-free survival among all and among resected patients with LAPC in the two arms in ITT | 60 months
  Comparison of overall and progression-free survival of patients with LAPC treated with standard or prolonged treatment. Comparison in survival will be performed among all enrolled patients and among all resected patients with LAPC receiving the two treatment durations
Overall/progression-free survival between all BR and LAPC patients in ITT | 60 months
  Comparison of overall/progression-free survival will be performed among all BR and LAPC patients - in the whole cohort, in the standard and in the prolonged treatment arm in ITT
Overall/progression-free survival between resected BR and LAPC patients in ITT | 60 months
  Comparison of overall/progression-free survival will be performed among resected BR and LAPC patients - in the whole cohort, in the standard and in the prolonged treatment arm in ITT
Resection rate | 24 months
  Difference in the proportion of resected patients (all and with BR and LAPC, respectively) between the standard and the prolonged NAT arm
N0 resection rate | 24 months
  Difference in the proportion of patients with no regional lymph node metastases (all and with BR and LAPC, respectively) between the standard and the prolonged NAT arm
90-day surgical complications | 12 months
  Difference in 90-days complication rates according to Clavien-Dindo among the resected patients treated in the standard and in the prolonged arms
Quality of life questionnaire EORTC QLQ-PAN26 | 60 months
  Comparison of quality of life evaluated by standardised questionnaires EORTC QLQ-PAN26 and PACADI between patients treated in the standard and the prolonged NAT group
Quality of life questionnaire PACADI | 60 months
  Comparison of quality of life evaluated by standardised questionnaire PACADI between patients treated in the standard and the prolonged NAT group
Biochemical response | 60 months
  Change in serum concentration of tumor markers CA19-9, CEA, CA125 before, during and after receipt of standard and prolonged NAT at specified time points
Chemotherapy start-rate and completion rate | 24 months
  Comparison of the proportion of patients who started and who completed NAT when receiving the standard and the prolonged NAT
Histopathologic response | 24 months
  Comparison of the proportion of patients who had the same grade of histopathologic tumor regression according to CAP when treated in the standard and in the prolonged NAT arms

CONTACTS AND LOCATIONS:
Overall Officials: Elena Rangelova, PhD, Principal Investigator — Sahlgrenska University Hospital, Västra Götalandsregion
Locations (1):
- SahlgrenskaUH, Gothenburg, VGR, Sweden